CLINICAL TRIAL: NCT00540371
Title: Dynamic Epidermal Cooling During Pulsed Dye Laser Treatment of Port Wine Stain
Brief Title: Dynamic Epidermal Cooling During Pulsed Dye Laser Treatment of Port Wine Stain Birthmark at High Fluences
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Kristen Kelly, M.D.,Professor Departments of Dermatology and Surgery, University of California, Irvine
Other Study IDs: 19992154
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Port Wine Stain
Keywords: Port Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Port wine stain Birthmark: Port wine stain Birthmark
  Interventions: Other: Port wine stain Birthmark

INTERVENTIONS:
Other: Port wine stain Birthmark — Port wine stain Birthmark

SUMMARY:
The purpose of the study is to improve the efficacy of pulsed dye laser treatment of port wine stain birthmarks. Involvement in the protocol will involve formal documentation of the level of treatment pain, duration of post-treatment purpura and incidence of side effects. In addition, measurements will be taken of blood substances that promote blood vessel formation/regrowth and non-invasive reflectance measurements and photographs will be taken before and after treatment.

The objective of this study is to document the degree of port wine stain lightening, the incidence of side effects and the presence of angiogenic factors induced during treatment with the pulsed dye laser in association with cooling agent. This information ultimately lead to improved treatment.

DETAILED DESCRIPTION:
The flashlamp-pumped pulsed dye laser has offered the best results with the lowest incidence of side effects. The yellow light is preferentially absorbed by hemoglobin allowing more selective destruction of the ectatic capillaries in the dermis.

The flashlamp-pumped pulsed dye laser has become the treatment of choice for port wine stain birthmarks; however, therapeutic challenges remain. The epidermis is not totally spared due to partial absorption of energy therein by melanin which presents an optical barrier through which the light must pass to reach the underlying blood vessels. Absorption of laser energy by melanin causes localized heating in the epidermis, which may, if not controlled, produce permanent complications such as hypertrophic scarring or dyspigmentation.

Clinical studies have demonstrated the efficacy and safety of cryogen spray cooling during pulsed laser treatment of port wine stain birthmarks. This technology allows the use of higher incident laser light dosages and has been demonstrated to improve treatment results. cryogen spray cooling also decreases treatment pain and the duration of post-laser treatment purpura.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PWS birthmark or age and sex matched control of a subject with a PWS birthmark
* Apparent good health as documented by medical history and physical examination
* Ability to understand and carry out subject instructions

Exclusion Criteria:

* Pregnancy
* History of cutaneous photosensitivity
* History of photodermatoses, skin cancer or other cancer
* Any therapy to the proposed treatment sites within the previous two months
* Current participation in any other investigational drug evaluation
* Concurrent use of known photosensitizing drugs
* Inability to understand and carry out subject instructions

Ages: 1 Month to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 1999-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Kelly, M.D, Principal Investigator — Beckman Laser Institue University of California Irvine
Locations (1):
- Beckman Lase Institute Medical Clinic Unversity of California Irvine, Irvine, California, United States